CLINICAL TRIAL: NCT01488916
Title: Impacts of Vitamin D Inadequacy on Postprandial Glucose Excursion in Patients With Type 2 Diabetes
Brief Title: Vitamin D Inadequacy on Postprandial Glucose in Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Principal Investgator, Taipei Veterans General Hospital, Taiwan
Other Study IDs: V100C-144-Protocol-1
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Type 2 Diabetes
Keywords: Vitamin D; Postprandial Glucose; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples after meal challenge
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Vitamin D deficiency: patients with serum vitamin D levels of the lower tertile
- Vitamin D inadequacy: patients with serum vitamin D levels of the middle tertile
- Reference group: patients with serum vitamin D levels of the upper tertile

SUMMARY:
Vitamin D deficiency is associated with an unfavorable metabolic profile in several observational studies. However, the influences of vitamin D concentrations on postprandial glucose in type 2 diabetes (DM) are less studied. The purposes of the study are to study the effects of vitamin D inadequacy on postprandial glucose excursion and metabolic responses in patients with type 2 DM. This is a cross-sectional study. About 150-180 patients will be screened for serum levels of 25(OH)D. A total of 45 eligible patients will be grouped into three groups by different vitamin D status: vitamin D deficiency, vitamin D insufficiency, and the controls. The patients will receive a mixed meal test for postprandial glucose excursion and metabolic responses. The investigators will use statistical methods to assess the differences in post-challenge glucose and metabolic response among the three groups of patients. The investigators hope the study can explore the relationship between vitamin D and glucose excursion in patients with type 2 DM.

DETAILED DESCRIPTION:
Vitamin D deficiency is associated with an unfavorable metabolic profile in several observational studies. However, the influences of vitamin D concentrations on postprandial glucose in type 2 diabetes (DM) are less studied. The purposes of the study are to study the effects of vitamin D inadequacy on postprandial glucose excursion and metabolic responses in patients with type 2 DM. This is a cross-sectional study. About 150-180 patients will be screened for serum levels of 25(OH)D. A total of 45 eligible patients will be grouped into three groups by different vitamin D status: vitamin D deficiency, vitamin D insufficiency, and the controls. The patients will receive a mixed meal test for postprandial glucose excursion and metabolic responses. Analysis of variance (ANOVA) will be applied to compare the differences in clinical characteristics among the three groups. Univariate analyses of general linear models will be used to compare the differences in meal-derived metabolic indexes among the three groups, showing effects of confounding variables including age, sex, obesity, and DM-related clinical parameters. Repeated-measures ANOVA will be used to assess the differences in post-challenge glucose and metabolic response in the meal test, with or without adjustments of the above covariates. Pearson and partial correlation procedures will be used to test the correlations of 25(OH)D with clinical parameters including lipid profile, HbA1c, and meal-derived metabolic indexes. Multiple linear regression models will be used in an attempt to compare the degree to which 25(OH)D concentrations is associated with the meal-derived metabolic indexes in these patients. The investigators hope the study can explore the relationship between vitamin D and glucose excursion in patients with type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory type 2 diabetes patients.
* Men or women.
* Aged 20 ~ 75 years old.
* Stable oral anti-diabetes therapy for at least 8 weeks.
* Willing to participate in the study by signing an informed consent.
* Willing to undergo a screening visit including medical history taking and fasting blood sampling.
* Willing to undergo a standardized mixed meal test at a separate visit.

Exclusion Criteria:

* Patients of type 2 diabetes with the following: History of HHNK; Fasting glucose higher than 250 mg/dL; Treated with insulin, alpha-glucosidase inhibitor, incretin mimetics, DPP-IV inhibitors or rapid-acting insulin secretagogus (the meglitinides) in the past 8 weeks;
* HbA1c > 8.5 %.
* History or evidence of parathyroid or calcium-related diseases.
* History or evidence of endocrine diseases including hyperthyroidism, hypothyroidism, adrenal disease and pituitary disease.
* History of major renal, liver, heart, blood and neurological disease, judged by the investigation physicians.
* History or evidence of alcoholism or drug abuse.
* History of surgical operation of upper gastrointestinal tract and liver. Women who are pregnant.
* History of malignancy within the last 5 years
* History of mental incapacity or language barriers that may preclude adequate understanding or cooperation in the study.
* Under systemic glucocorticoid therapy in the past 8 weeks
* Under supplementation of vitamin D, of any kind, in the past 4 weeks
* Under hormonal replacement therapy in the past 8 weeks
* Under treatments for osteoporosis including calcitonin and biphosphate in the past 8 weeks.
* History or evidence of difficult venous access
* Subjects with the following laboratory values: hemoglobin < 9 g/dL, WBC < 3000/mL, platelet < 100,000/mL, serum Cr > 2.0 mg/dL, ALT > 3x ULN, total bilirubin > 2x ULN.
* Current or concomitant illness that would interfere with the subject's ability to perform the study or that would confound the study results, judged by the investigation physicians.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the present study, we propose to screen patients with type 2 DM for vatamin D inadequacy. Those with different vitamin D status will be invited to participate in a mixed meal test.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
incremental areas under the curves of plasma glucose after meal challenge | 20 days
  Within 20 days of the screening visit, the eligible participants will receive a 3-h mixed meal test for postprandial glucose excursion.

SECONDARY OUTCOMES:
insulin sensitivity and β-cell function indexes from the meal test | 20 days
  Within 20 days of the screening visit, the eligible participants will receive a 3-h mixed meal test for postprandial glucose excursion.
Meal-related glycemic excursion indexes (∆G, ∆T, BR)from the meal test | 20 days
  Within 20 days of the screening visit, the eligible participants will receive a 3-h mixed meal test for postprandial glucose excursion.

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Min Hwu, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan